CLINICAL TRIAL: NCT05689515
Title: PL4Y: A Pilot Randomized Control Trial to Study the Feasibility of Positive Links for Youth Care Engagement Intervention
Brief Title: Feasibility of Positive Links for Youth Care Engagement Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC20220752H; 5R34MH122332-03 (NIH)
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: HIV Antibody Positivity
Keywords: Positive Links; Youth; Emerging Adults
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:1 ratio to intervention (PL4Y use) or standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Health App group (Experimental): Mobile health app to increase rates of engagement in care in youths living with HIV
  Interventions: Behavioral: Mobile health app
- Control group (No Intervention): Standard of care for youths living with HIV

INTERVENTIONS:
Behavioral: Mobile health app — A mobile app provided to participants to assess effectiveness in managing HIV
  Other Names: PL4Y
  Arms: Mobile Health App group

SUMMARY:
A small pilot study to assess feasibility and acceptability of the PL4Y intervention.

DETAILED DESCRIPTION:
After completing enrollment and informed consent, participants will be randomly assigned to PL4Y in a 2:1 fashion (intervention:control) with a target enrollment of 40 receiving the intervention and 20 in the control arm for a total of 60 participants. There is no blinding in this study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection
* Recent diagnosis of HIV (within the past 6 months) OR be virologically unsuppressed (>1000 copies/ml) OR disengaged from HIV care (< 2 visits/last 12 months > 90 days apart)

Exclusion Criteria:

* Cannot consent
* Unwilling to come to visits
* Unwilling to be in San Antonio for a year

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Completion of Feasibility Survey | 12 months
  Feasibility survey completion by participants regarding usability of the PL4Y intervention
Viral plasma load measurement | 12 months
  Virologic suppression is the primary goal of HIV treatment. Virologic failure is defined as a measurement over 200 copies per mL by the Department of Health and Human Services, and is the primary determinant of successful HIV control.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Taylor, MD, MS, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University Health Center Downtown, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will compose a manuscript including data on preliminary efficacy of the PL4Y program in YLWH with regards to virologic suppression, retention in care, stigma, self-efficacy, and social support. The study team will also have a detailed guide to operating procedures, including successful recruitment and retention techniques and study processes such as teching tarticipants how to use PL4Y and monitoring the community message board. All data regarding participants will be shared as de-identified data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At study completion and when all data have been analyzed to publish in a peer reviewed journal.

DOCUMENTS (1):
  • Informed Consent Form (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT05689515/ICF_000.pdf